CLINICAL TRIAL: NCT02681042
Title: Left Atrial Appendage Closure With SentreHeart Lariat® Device
Acronym: Lariat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 014-292
Record Dates: First submitted 2015-05-26; First posted 2016-02-12 (Estimated); Results first posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Cardioembolic Stroke; Atrial Fibrillation
MeSH Terms: conditions — Embolic Stroke; Atrial Fibrillation | interventions — Left Atrial Appendage Closure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SentreHeart Lariat (Experimental): Left atrial appendage closure with SentreHeart Lariat device
  Interventions: Procedure: Left atrial appendage closure; Device: SentreHeart Lariat®

INTERVENTIONS:
Procedure: Left atrial appendage closure — The SentreHeart Lariat® device (that is approved for soft tissue ligation) will be used to ligate or close the left atrial appendage as a stand-alone procedure at the participating centers.
Device: SentreHeart Lariat® — The SentreHeart Lariat® device (that is approved for soft tissue ligation) will be used to ligate or close the left atrial appendage as a stand-alone procedure at the participating centers.

SUMMARY:
The study cohort will consist of up to 50 patients who are candidates for Left Atrial Appendage (LAA) closure in whom oral anticoagulation is contraindicated.

Subjects evaluated for left atrial appendage closure will be screened for inclusion and consented prior to their procedure. If the anatomy is favorable for placement of the Lariat® device, the procedure will be performed at one of the participating centers. If anatomy is not favorable, the patient will be excluded from the study and managed using best care practices by his or her physician.

DETAILED DESCRIPTION:
The study cohort will consist of up to 50 patients who are candidates for LAA closure in whom oral anticoagulation is contraindicated.

Subjects evaluated for left atrial appendage closure will be screened for inclusion and consented prior to their procedure. If the anatomy is favorable for placement of the Lariat® device, the procedure will be performed at one of the participating centers. If anatomy is not favorable, the patient will be excluded from the study and managed using best care practices by his or her physician.

Subjects consented will be tracked by the study team and will be considered enrolled in this study at the time of the start of their left atrial appendage closure procedure. All subjects that are consented who do not undergo left atrial appendage closure with SentreHeart Lariat® will be considered screen failures. Any patients that have a failed attempt at left atrial appendage closure with SentreHeart Lariat® will be tracked through their index hospitalization for safety; their study follow up will be complete at the time of discharge.

The invasive procedure for placement of the study devices will proceed according to standard interventional techniques, as already in place at the participating centers. Patients undergoing the Lariat® procedure will be administered colchicine 0.6 mg po twice daily for a minimum of three days preoperatively, and 30 days postoperatively. (This dose may be adjusted for renal function or intolerance).

Patients will undergo follow-up visits at 7 days, 90 days, and 180 days post procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years
* Patients able and willing to provide informed consent
* Documentation of atrial fibrillation or atrial flutter
* Clinical decision by the subject's physician that the patient is at risk for embolic stroke, and oral anticoagulant medications (OAC) is contraindicated
* Hypertension, Abnormal renal and hepatic function, Stroke, Bleeding tendency/predisposition, Labile International Normalized Ratios (INRs) on warfarin (HAS-BLED) score > 3
* Congestive Heart Failure (CHF), Hypertension, Age >65, Diabetes Mellitus, Stroke or Transient Ischemic Attack (TIA), Vascular Disease, Age >75, Sex Category (CHADS2-VASC) score >3, OR CHADS2-VASC of 2 if physician provides justification for procedure
* Anatomy favorable for deployment of the SentreHeart Lariat®

Exclusion Criteria:

* Medically unable to provide informed consent
* Previous cardiothoracic surgery
* Patient is a candidate for catheter or surgical ablation
* Need for concomitant cardiac surgery procedure
* Thrombus in the left atrial appendage or left atrium
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2018-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. B. DeVille, MD, Principal Investigator — Prinicpal Investigator
Locations (1):
- Baylor Research Institute at The Heart Hospital Baylor Plano, Plano, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 4 different hospitals.
Pre-assignment Details: Patients were enrolled, but if the implant of the Lariat device was not successful, patients would be exited from the trial. All patients with successful implant were followed for 180 days.
Period: Overall Study
Arm/Group | SentreHeart Lariat
Started | 9
Completed | 6
Not Completed | 3
Not completed — Implant Failure | 3

BASELINE CHARACTERISTICS:
Population: 9 patients were enrolled and had the the Sentreheart device implantation attempted
Arm/Group | SentreHeart Lariat
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 7
Age, Continuous [Mean (Full Range); unit: years] | 73.6 [58 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Stand-Alone Left Atrial Appendage Closure Using SentreHeart Lariat Device as Measured by Left Atrial Appendage Closure Rates
Description: The primary aim is to assess the outcome of patients undergoing left atrial appendage ligation or closure with the SentreHeart Lariat® device as a stand-alone procedure at the participating centers
Time Frame: 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | SentreHeart Lariat
Number analyzed (Participants) | 9
Participants | 6

2. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: Secondary aims include assessment of adverse events
Time Frame: 180 days
Measure: Number; unit: patients with adverse events
Arm/Group | SentreHeart Lariat
Number analyzed (Participants) | 9
patients with adverse events | 6

3. Secondary Outcome: Successful LAA Closure Rate
Description: Secondary aims include successful LAA closure rates
Time Frame: 180 days
Population: Number of patients with successful left atrial appendage closure
Measure: Count of Participants; unit: Participants
Arm/Group | SentreHeart Lariat
Number analyzed (Participants) | 9
Participants | 6

ADVERSE EVENTS:
Time Frame: 180 days
Description: Adverse events were collected as standard
Arm/Group | SentreHeart Lariat
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 2/9
Other Adverse Events (participants affected / at risk) | 6/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SentreHeart Lariat (N=9)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Positive nuclear stress test (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SentreHeart Lariat (N=9)
hypotension (Cardiac disorders) | 2 (2) — hypotension
diarrhea (Gastrointestinal disorders) | 1 (1) — diarrhea
UTI (Renal and urinary disorders) | 1 (1) — Urinary Tract Infection
pericardial effusion (Cardiac disorders) | 1 (1) — microtear pericardial effusion
unspecified chest pain (Cardiac disorders) | 1 (1) — unspecified chest pain
bilateral pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) — bilateral pleural effusion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-06-08): https://cdn.clinicaltrials.gov/large-docs/42/NCT02681042/Prot_SAP_000.pdf
  • Informed Consent Form (2016-09-27): https://cdn.clinicaltrials.gov/large-docs/42/NCT02681042/ICF_001.pdf